CLINICAL TRIAL: NCT00199914
Title: The Effectiveness of Shortwave Diathermy in Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Efficacy Study of Shortwave Diathermy for the Treatment of Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Rattanachaiyanont, M.D., Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34/2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee; Menopause
Keywords: Diathermy; Short-wave therapy; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Fever; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The treatment group received short-wave diathermy (SWD) plus exercise whereas the control group received exercise alone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shortwave diathermy (Experimental): continuous shortwave diathermy, 20 min/session, 3 sessions/week for 3 weeks
  Interventions: Device: Shortwave diathermy
- control (Sham Comparator): continuous sham shortwave diathermy, 20 min/session, 3 sessions/week for 3 weeks
  Interventions: Device: Shortwave diathermy

INTERVENTIONS:
Device: Shortwave diathermy — continuous shortwave diathermy, 20 min/session, 3 sessions/week for 3 weeks

SUMMARY:
The purpose of this study is to determine whether shortwave diathermy is effective in reducing knee pain and increasing function of the patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common degenerative joint disease, resulting in significant morbidity and health care expense. It affects more than 60% of Western World adults over the age of 65 years. It causes pain and dysfunction in 20% of elderly persons. It can affect any joint containing hyaline cartilage; knee is the most commonly affected joint. There are many strategies for the treatment of knee OA but a curative method has not been found. Treatment is therefore aimed to relief symptoms and to prevent further functional deterioration. It is unclear whether any of the treatment modalities is efficacious. Shortwave diathermy (SWD) is one of deep heat widely applied to alleviate the symptoms associated with OA. The efficacy of SWD for the treatment of OA knee is still inconclusive. The outcome of treatment in previous reports varies from null to positive effect. This discrepancy is largely due to the different research methodology, the inadequate sample size, the methods used in outcome assessment, and the treatment protocols.

Comparison(s): Peri- or postmenopausal women with OA knee are randomized into two groups, receiving a course of either therapeutic SWD or sham SWD. The main outcome measured is the change in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index.

ELIGIBILITY:
Inclusion Criteria:

* peri- or postmenopausal women aged >50 years
* primary knee osteoarthritis

Exclusion Criteria:

* inability to walk
* severe joint instability
* history of previous shortwave diathermy
* intra-articular injection within 3 months
* metallic implant around knee joint
* suspicious of malignancy around knee joint
* significant cardiovascular disease
* inability to understand how to score the symptoms

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-01; Primary Completion 2004-05 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manee Rattanachaiyanont, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The present study start date was before January 18, 2017; therefore we did not plan to share IPD. However, the IPD is available upon request to the correspondent.

REFERENCES:
- [Result] Rattanachaiyanont M, Kuptniratsaikul V. No additional benefit of shortwave diathermy over exercise program for knee osteoarthritis in peri-/post-menopausal women: an equivalence trial. Osteoarthritis Cartilage. 2008 Jul;16(7):823-8. doi: 10.1016/j.joca.2007.10.013. Epub 2008 Feb 21. PMID 18178111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized and double blind placebo controlled equivalence trial was carried out in the out-patient clinic, Department of Rehabilitation Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University from January to June 2004.
Pre-assignment Details: All patients had primary knee OA and without the following conditions: inability to walk, severe joint instability, history of previous SWD treatment, intra-articular injection within 3 months, metallic implant around knee joint, suspicious of malignancy around knee joint, significant cardiovascular disease.
Period: Overall Study
Arm/Group | Shortwave Diathermy | Control
Started | 53 | 60
Completed | 50 | 54
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shortwave Diathermy | Control | Total
Number analyzed (Participants) | 53 | 60 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.32 (7.61) | 62.48 (8.47) | 62.88 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 60 | 113
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 53 | 60 | 113

OUTCOME MEASURES:

1. Primary Outcome: The Change in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index
Description: The WOMAC index is a multidimensional, self-administered health status evaluation instrument for patients with OA of the hip and knee. It is composed of 24 items that are grouped into three dimensions, including pain (5 items), stiffness (2 items), and function (17 items). The response can be in a form of visual analog or five-point Likert scale [11, 23]. In this study, the response is on a 10-cm horizontal line with numeric description from 0 to 10. The score of each dimension is an average of the component item scores. The WOMAC total score is determined by averaging the scores of all dimensions. The total score ranges from 0 (best outcome possible) to 10 (worst outcome possible).
Time Frame: 3 weeks
Population: Statistical analyses to test the superiority were based on the intention-to-treat (ITT) population, and those chosen to demonstrate the equivalence were based on the per protocol population. The "worst -case-scenario" was applied to the dropouts in the ITT analyses.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shortwave Diathermy | Control
Number analyzed (Participants) | 54 | 60
units on a scale | 0.71 [0.42 to 0.99] | 0.65 [0.37 to 0.92]

2. Secondary Outcome: Gait Speed (Calculated From the Time Spending for 100-meter Walk)
Time Frame: 3 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Global Improvement
Time Frame: 3 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Patient's Satisfaction to the Treatment
Time Frame: 3 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Adverse Events
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Shortwave Diathermy | Control
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 4/50 | 4/54
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shortwave Diathermy (N=50) | Control (N=54)
pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
flushing (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The present study has limitations in generalizability. The study population was peri-/post-menopausal Thai women whose lifestyle might be different from that of other ethnic groups. The relatively short duration of treatment might not be sufficient to show the benefit of short-wave diathermy (SWD) treatment. Only one SWD machine with a unique output power was used in order to homogenize the provided treatment. All of these conditions would make the results in-applicable to different situations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes